CLINICAL TRIAL: NCT00065377
Title: An Exploratory Study of the Effects of Oral Glucosamine Administration on Insulin Sensitivity and Capillary Recruitment in Normal and Obese Subjects
Brief Title: Effects of Oral Glucosamine on Insulin and Blood Vessel Activity in Normal and Obese People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030251; 03-AT-0251
Record Dates: First submitted 2003-07-21; First posted 2003-07-22 (Estimated); Last update posted 2006-06-26 (Estimated); Status verified 2006-06

CONDITIONS: Obesity; Insulin Resistance
Keywords: Diabetes; Insulin Resistance; Capillary Blood Flow; Osteoarthritis; Endothelial Dysfunction; Obesity; Healthy Volunteer; HV
MeSH Terms: conditions — Obesity; Insulin Resistance; Diabetes Mellitus; Osteoarthritis | interventions — Glucosamine

INTERVENTIONS:
Drug: Glucosamine Hydrochloride

SUMMARY:
This study will examine whether glucosamine affects the way the body responds to insulin. Insulin is a hormone that causes the body to use glucose (sugar). Insulin does not work as well in overweight people, causing a condition called insulin resistance. Insulin also increases the flow of blood into muscle by opening inactive blood vessels. This study will test whether glucosamine, a nutritional supplement that many people take to treat arthritis, can cause or worsen insulin resistance or change how blood vessels react to insulin in normal weight and overweight people.

Healthy normal weight and overweight volunteers between 21 and 65 years of age may be eligible for this study. Candidates will be screened with a brief physical examination, medical history, and blood and urine tests. After screening, participants will have three additional outpatient clinic visits for the following procedures:

Visit 1

* Glucose clamp test to measure the body's response to insulin: For this procedure, a needle is placed in a vein of each arm, one for drawing blood samples, and one for infusing glucose and a potassium solution. The glucose is infused continuously during this 4-hour test and blood is drawn frequently to monitor glucose and insulin levels. After the test, blood glucose levels are monitored for another 2 hours to make sure they remain at an adequate level to prevent hypoglycemia (low blood sugar).
* Blood flow measurement: Blood flow in the brachial artery of the arm is measured to assess how many capillaries (very small blood vessels) are being used to supply nutrients and oxygen to the muscle in the forearm. This test is done at the same time as the glucose clamp test. Blood flow is measured using a technique called contrast ultrasound. A small amount of contrast agent consisting of gas-filled bubbles the size of red blood cells is infused over 10 minutes through one of the catheters placed in the vein for the glucose clamp test. The contrast agent is infused twice, once at the beginning of the glucose clamp test and once at the end of the test. The contrast material creates a signal in response to ultrasound that provides information about the distribution of capillaries in the forearm.
* Assignment to medication group: Participants are randomly assigned to take either glucosamine or placebo three times a day by mouth for 6 weeks. At the end of the 6 weeks, no study drug is taken for 1 week, and then participants "cross-over" medications, those who took glucosamine for the first 6 weeks take placebo for the next 6 weeks and vice versa.

Visits 2 and 3

For these visits, the glucose clamp test and blood flow measurements are repeated. Visit 2 is scheduled at the end of the first 6-week treatment period, and Visit 3 is scheduled at the end of the second 6-week treatment period.

DETAILED DESCRIPTION:
Glucosamine is a popular over-the-counter nutritional supplement that many people use for the treatment of osteoarthritis. Intravenous administration of glucosamine to animals or humans causes significant metabolic insulin resistance and vascular endothelial dysfunction. Moreover, experiments with various cell lines have implicated elevated glucosamine levels in the development of insulin resistance. However, there are no published studies examining the potential effects of oral glucosamine administration to modulate insulin sensitivity or capillary recruitment in humans. This is a significant concern because insulin resistance and vascular dysfunction contribute importantly to major public health problems including diabetes, obesity, hypertension, and cardiovascular diseases. Normal healthy volunteers and obese insulin resistant subjects will be enrolled in a randomized double-blind, placebo-controlled, crossover study to evaluate the effects of oral glucosamine to modulate insulin sensitivity and insulin-stimulated capillary recruitment. The reference standard hyperinsulinemic isoglycemic glucose clamp technique will be used to assess insulin sensitivity before treatment, after placebo or oral glucosamine (500 mg p.o. TID for 6 weeks), and after completion of the crossover. In addition, insulin-stimulated capillary recruitment will be measured at the same time as the glucose clamp studies by using the ultrasound microbubble contrast technique to assess blood flow in the brachial artery and capillary recruitment in forearm skeletal muscle in response to hyperinsulinemia. Finally, plasma glucosamine levels will be measured just prior to each glucose clamp study using an HPLC method. The results of this study will determine if oral glucosamine administration causes significant insulin resistance and impairment in insulin-stimulated capillary recruitment in healthy volunteers or worsens insulin resistance and capillary recruitment in obese subjects. In addition, our study will provide important information about how plasma glucosamine levels change with commonly used oral doses of glucosamine.

ELIGIBILITY:
* INCLUSION CRITERIA:

HEALTHY VOLUNTEERS:

Males or females in good general health with no significant underlying illnesses, on no medication, between the ages of 21-65 years of age with HbA1C less than 6.5, fasting blood glucose less than 100 mg/dl, blood pressure less than 130/85, and BMI between 20-26 kg/m(2). Subjects should have never smoked tobacco or not smoked within the previous 2 years.

OBESE SUBJECTS:

Males or females in good general health with no significant underlying illnesses, on no medication, between the ages of 21-65 years of age with HbA1C less than 6.5, fasting blood glucose less than 110 mg/dl, blood pressure less than 130/85, and BMI between 30-40 kg/m(2).

EXCLUSION CRITERIA:

Subjects will be excluded if they have diabetes, hypertension, pregnancy, liver disease, pulmonary disease, renal insufficiency, coronary heart disease, heart failure, peripheral vascular disease, coagulopathy, actively smoking within last two years, in treatment for any form of cancer, positive tests for HIV, hepatitis B or C, or take systemic corticosteroids.

Subjects will also be excluded if they have an allergy to shellfish since glucosamine is derived from shellfish. Subjects will be excluded if they have taken glucosamine within the last three months. Subjects with allergies to blood products or eggs or known hypersensitivity to albumin will also be excluded from participating because of potential adverse effects from microbubble contrast agent. Subjects will be excluded from this study because children do not typically take glucosamine or have osteoarthritis.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-07; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Center for Complementary and Alternative Medicine (NCCAM), Bethesda, Maryland, United States

REFERENCES:
- [Background] Barclay TS, Tsourounis C, McCart GM. Glucosamine. Ann Pharmacother. 1998 May;32(5):574-9. doi: 10.1345/aph.17235. PMID 9606479
- [Derived] Muniyappa R, Karne RJ, Hall G, Crandon SK, Bronstein JA, Ver MR, Hortin GL, Quon MJ. Oral glucosamine for 6 weeks at standard doses does not cause or worsen insulin resistance or endothelial dysfunction in lean or obese subjects. Diabetes. 2006 Nov;55(11):3142-50. doi: 10.2337/db06-0714. PMID 17065354